CLINICAL TRIAL: NCT01154270
Title: Combined Therapy of Malignant Salivary Gland Tumours With IMRT and Carbon Ions: COSMIC
Brief Title: CO(Mbined Therapy of Malignant) S(Alivary Gland tu)M(Ours With)I(MRT and) c(Arbon Ions): COSMIC
Acronym: COSMIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: PD Dr. MW Münter, Dept. of Radiation Oncology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COSMIC
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Malignancy; Salivary Glands; Tumor
Keywords: cancer of the salivary glands; radiation; carbon ion therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT + C12-boost (Experimental): (8 x 3 GyE) carbon ion therapy followed by 50 Gy IMRT (2 Gy/ Fx)corresponding to a total dose of approximately 74 GyE.
  Interventions: Radiation: carbon ion boost

INTERVENTIONS:
Radiation: carbon ion boost — 8 fractions carbon ion (8 x 3 GyE C12) therapy followed by 25 fractions of IMRT corresponding to a total dose of approximately 74 GyE. Treatment duration is approximately 61/2-7 weeks

SUMMARY:
The COSMIC trial is a prospective, mono-centric, phase II trial evaluating toxicity and efficacy in the combined treatment with intensity-modulated radiation therapy (IMRT) and carbon ion (C12) boost. Primary endpoint is mucositis ≥ CTC°3, secondary endpoints are local control, disease-free survival, and toxicity. Planned accrual of the trial includes 54 patients with histologically proved (≥R1-resected, inoperable or Pn+) salivary gland malignancies. Treatment consists of 24 GyE carbon ions (8 fractions) and 50 Gy IMRT (2.0 Gy/ fraction).

DETAILED DESCRIPTION:
Local control in malignant salivary gland tumours is dose dependent. High local control rates in adenoid cystic carcinomas could be achieved by highly conformal radiotherapy techniques and particle (neutron/ carbon ion) therapy. Considering high doses are needed to achieve local control, all malignant salivary gland tumours probably profit from the use of particle therapy, which in case of carbon ion treatment, has been shown to be accompanied by only mild side-effects.

Methods/ design:

The COSMIC trial is a prospective, mono-centric, phase II trial evaluating toxicity in the combined treatment with intensity-modulated radiation therapy (IMRT) and carbon ion (C12) boost in 54 patients with histologically proved (≥R1-resected, inoperable or Pn+) salivary gland malignancies. Patients receive 24 GyE carbon ions (8 fractions) and IMRT (2.0 Gy/ fraction).

Study objectives:

Incidence of mucositis ≥ CTC°3 will be assessed as the primary endpoint of the trial, local control, disease-free survival, toxicity (incl. mucositis CTC °I-II and late toxicity at 3 years post RT)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or surgically removed malignant tumour of the salivary glands (head and neck)
* Inoperable tumour
* G2/3
* Macroscopic or microscopic residual tumour (R2/ R1) or
* ≥T3/T4 or
* perineural invasion (Pn+)
* written informed consent
* pts aged 18 - 80 years
* effective contraception for pts in childbearing age (<12 months post beginning of menopause)

Exclusion Criteria:

* Prior radio- or chemotherapy for tumours of the head and neck
* Other previous malignancy within the past 5 years except prior, adequately treated basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Significant neurological or psychiatric condition including dementia or seizures or other serious medical condition prohibiting the patient's participation in the trial by judgement of the investigators
* Legal incapacity or limited legal capacity
* Positive serum/ urine beta-HCG/ pregnancy
* Drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
mucositis ≥ CTC°3 | 6-8 weeks post completion of treatment

SECONDARY OUTCOMES:
local control | 3 years post RT
  to evaluate local control at 3 years post RT
acute toxicity | 6-8 weeks post completion of treatment
  evaluation of acute radiation effects (other than mucositis CTC°C) 6-8 weeks post completion of treatment
late toxicity | 3 years post radiotherapy
  to evaluate radiation late effects
disease-free survival | 3 years post treatment
  to evaluate disease-free survival at 3 years post radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc W Muenter, MD, Principal Investigator — Dept. of Radiation Oncology, INF 400, 69120 Heidelberg
Locations (1):
- Dept. of Radiation Oncology, INF 400, Heidelberg, Germany

REFERENCES:
- [Background] Spiro RH. Salivary neoplasms: overview of a 35-year experience with 2,807 patients. Head Neck Surg. 1986 Jan-Feb;8(3):177-84. doi: 10.1002/hed.2890080309. PMID 3744850
- [Background] Chen AM, Granchi PJ, Garcia J, Bucci MK, Fu KK, Eisele DW. Local-regional recurrence after surgery without postoperative irradiation for carcinomas of the major salivary glands: implications for adjuvant therapy. Int J Radiat Oncol Biol Phys. 2007 Mar 15;67(4):982-7. doi: 10.1016/j.ijrobp.2006.10.043. Epub 2007 Jan 22. PMID 17241753
- [Background] Gurney TA, Eisele DW, Weinberg V, Shin E, Lee N. Adenoid cystic carcinoma of the major salivary glands treated with surgery and radiation. Laryngoscope. 2005 Jul;115(7):1278-82. doi: 10.1097/01.MLG.0000165381.64157.AD. PMID 15995521
- [Background] Mendenhall WM, Morris CG, Amdur RJ, Werning JW, Hinerman RW, Villaret DB. Radiotherapy alone or combined with surgery for adenoid cystic carcinoma of the head and neck. Head Neck. 2004 Feb;26(2):154-62. doi: 10.1002/hed.10380. PMID 14762884
- [Background] Chen AM, Bucci MK, Weinberg V, Garcia J, Quivey JM, Schechter NR, Phillips TL, Fu KK, Eisele DW. Adenoid cystic carcinoma of the head and neck treated by surgery with or without postoperative radiation therapy: prognostic features of recurrence. Int J Radiat Oncol Biol Phys. 2006 Sep 1;66(1):152-9. doi: 10.1016/j.ijrobp.2006.04.014. PMID 16904520
- [Background] Garden AS, Weber RS, Ang KK, Morrison WH, Matre J, Peters LJ. Postoperative radiation therapy for malignant tumors of minor salivary glands. Outcome and patterns of failure. Cancer. 1994 May 15;73(10):2563-9. doi: 10.1002/1097-0142(19940515)73:103.0.co;2-x. PMID 8174054
- [Background] Terhaard CH, Lubsen H, Van der Tweel I, Hilgers FJ, Eijkenboom WM, Marres HA, Tjho-Heslinga RE, de Jong JM, Roodenburg JL; Dutch Head and Neck Oncology Cooperative Group. Salivary gland carcinoma: independent prognostic factors for locoregional control, distant metastases, and overall survival: results of the Dutch head and neck oncology cooperative group. Head Neck. 2004 Aug;26(8):681-92; discussion 692-3. doi: 10.1002/hed.10400. PMID 15287035
- [Background] Terhaard CH, Lubsen H, Rasch CR, Levendag PC, Kaanders HH, Tjho-Heslinga RE, van Den Ende PL, Burlage F; Dutch Head and Neck Oncology Cooperative Group. The role of radiotherapy in the treatment of malignant salivary gland tumors. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):103-11. doi: 10.1016/j.ijrobp.2004.03.018. PMID 15629600
- [Background] Bittner N, Koh WJ, Laramore GE, Patel S, Mulligan MS, Douglas JG. Treatment of locally advanced adenoid cystic carcinoma of the trachea with neutron radiotherapy. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):410-4. doi: 10.1016/j.ijrobp.2008.01.016. Epub 2008 Apr 18. PMID 18374509
- [Background] Schulz-Ertner D, Nikoghosyan A, Didinger B, Munter M, Jakel O, Karger CP, Debus J. Therapy strategies for locally advanced adenoid cystic carcinomas using modern radiation therapy techniques. Cancer. 2005 Jul 15;104(2):338-44. doi: 10.1002/cncr.21158. PMID 15937907
- [Background] Douglas JG, Koh WJ, Austin-Seymour M, Laramore GE. Treatment of salivary gland neoplasms with fast neutron radiotherapy. Arch Otolaryngol Head Neck Surg. 2003 Sep;129(9):944-8. doi: 10.1001/archotol.129.9.944. PMID 12975266
- [Background] Mizoe JE, Tsujii H, Kamada T, Matsuoka Y, Tsuji H, Osaka Y, Hasegawa A, Yamamoto N, Ebihara S, Konno A; Organizing Committee for the Working Group for Head-And-Neck Cancer. Dose escalation study of carbon ion radiotherapy for locally advanced head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2004 Oct 1;60(2):358-64. doi: 10.1016/j.ijrobp.2004.02.067. PMID 15380567
- [Background] Huber PE, Debus J, Latz D, Zierhut D, Bischof M, Wannenmacher M, Engenhart-Cabillic R. Radiotherapy for advanced adenoid cystic carcinoma: neutrons, photons or mixed beam? Radiother Oncol. 2001 May;59(2):161-7. doi: 10.1016/s0167-8140(00)00273-5. PMID 11325445
- [Background] Munter MW, Schulz-Ertner D, Hof H, Nikoghosyan A, Jensen A, Nill S, Huber P, Debus J. Inverse planned stereotactic intensity modulated radiotherapy (IMRT) in the treatment of incompletely and completely resected adenoid cystic carcinomas of the head and neck: initial clinical results and toxicity of treatment. Radiat Oncol. 2006 Jun 6;1:17. doi: 10.1186/1748-717X-1-17. PMID 16756669
- [Background] Pommier P, Liebsch NJ, Deschler DG, Lin DT, McIntyre JF, Barker FG 2nd, Adams JA, Lopes VV, Varvares M, Loeffler JS, Chan AW. Proton beam radiation therapy for skull base adenoid cystic carcinoma. Arch Otolaryngol Head Neck Surg. 2006 Nov;132(11):1242-9. doi: 10.1001/archotol.132.11.1242. PMID 17116822
- [Background] Schulz-Ertner D, Nikoghosyan A, Jakel O, Haberer T, Kraft G, Scholz M, Wannenmacher M, Debus J. Feasibility and toxicity of combined photon and carbon ion radiotherapy for locally advanced adenoid cystic carcinomas. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):391-8. doi: 10.1016/s0360-3016(02)04511-x. PMID 12738314
- [Background] Schulz-Ertner D, Nikoghosyan A, Thilmann C, Haberer T, Jakel O, Karger C, Kraft G, Wannenmacher M, Debus J. Results of carbon ion radiotherapy in 152 patients. Int J Radiat Oncol Biol Phys. 2004 Feb 1;58(2):631-40. doi: 10.1016/j.ijrobp.2003.09.041. PMID 14751537
- [Background] Münter M, Umathum V, Nikoghosyan A, Jensen A, Hof H, Jaekel O, et al. Combination of intensity modulated radiation therapy (IMRT) and a carbon ion boost for subtotal resected or inoperable adenoid cystic carcinomas (ACC's) of the head and neck. PTCOG meeting 2009, abstract FC84
- [Background] Krempien R, Münter MW, Timke C, Friess H, Hartung G, Herfarth KK, et al. Cetuximab in combination with intensity modulated radiotherapy (IMRT) and gemcitabine for patients with locally advanced pancreatic cancer: a prospective phase II trial [PARC-study ISRCTN56652283]. J Clin Oncol 2007; 25 (18S) 4573
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Derived] Jensen AD, Nikoghosyan AV, Lossner K, Herfarth KK, Debus J, Munter MW. IMRT and carbon ion boost for malignant salivary gland tumors: interim analysis of the COSMIC trial. BMC Cancer. 2012 May 2;12:163. doi: 10.1186/1471-2407-12-163. PMID 22551422
- [Derived] Jensen AD, Nikoghosyan A, Windemuth-Kieselbach C, Debus J, Munter MW. Combined treatment of malignant salivary gland tumours with intensity-modulated radiation therapy (IMRT) and carbon ions: COSMIC. BMC Cancer. 2010 Oct 11;10:546. doi: 10.1186/1471-2407-10-546. PMID 20937120